CLINICAL TRIAL: NCT05245552
Title: An Open Phase I and Randomized, Double-blind, Controlled Phase III Clinical Trial to Evaluate the Safety and Immunogenicity of Quadrivalent Influenza Vaccine in Healthy Subjects Aged 6 to 35months.
Brief Title: A Clinical Trial of Quadrivalent Influenza Vaccine in Healthy Subjects Aged 6 to 35 Months
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PRO-QINF-3003
Record Dates: First submitted 2022-02-08; First posted 2022-02-18 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Seasonal Influenza
MeSH Terms: interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Safety group (Experimental): PhaseⅠ,30 subjects will receive two doses of quadrivalent influenza vaccine(0.5ml) on the immunization schedule of day 0,28.
  Interventions: Biological: Quadrivalent influenza vaccine(0.25ml)
- Experimental Group of quadrivalent influenza vaccine(0.25ml) (Experimental): 1100 subjects phase III will receive two doses of quadrivalent influenza vaccine(0.25ml) on the immunization schedule of day 0,28.
  Interventions: Biological: Quadrivalent influenza vaccine(0.25ml)
- Experimental Group of quadrivalent influenza vaccine(0.5ml) (Experimental): 1100 subjects phase III will receive two doses of quadrivalent influenza vaccine(0.5ml) on the immunization schedule of day 0,28.
  Interventions: Biological: Quadrivalent influenza vaccine(0.5ml)
- Control Group of trivalent influenza vaccine(BV) (Active Comparator): 550 subjects phase III will receive two doses of trivalent influenza vaccine(BV) on the immunization schedule of day 0,28.
  Interventions: Biological: Trivalent influenza vaccine(BV)
- Control Group of trivalent influenza vaccine(BY) (Active Comparator): 550 subjects phase III will receive two doses of trivalent influenza vaccine(BY) on the immunization schedule of day 0,28.
  Interventions: Biological: Trivalent influenza vaccine(BY)

INTERVENTIONS:
Biological: Quadrivalent influenza vaccine(0.25ml) — 7.5 ug hemagglutinin (HA) of each of the four influenza strains in 0.25 mL of sodium chloride, disodium hydrogen phosphate, sodium dihydrogen phosphate per injection.The routine of administration is Intramuscular injection into deltoid region.And the immunization schedule is two doses of quadrivalent influenza vaccine on day 0, 28.
  Arms: Experimental Group of quadrivalent influenza vaccine(0.25ml); Safety group
Biological: Quadrivalent influenza vaccine(0.5ml) — 15 ug hemagglutinin (HA) of each of the four influenza strains in 0.5 mL of sodium chloride, disodium hydrogen phosphate, sodium dihydrogen phosphate per injection.The routine of administration is Intramuscular injection into deltoid region.And the immunization schedule is two doses of quadrivalent influenza vaccine on day 0, 28.
  Arms: Experimental Group of quadrivalent influenza vaccine(0.5ml)
Biological: Trivalent influenza vaccine(BV) — 7.5μg inactivated influenza antigen (H1N1, H3N2, Victoria) of each of the trivalent influenza vaccine in 0.25 mL of sodium chloride, disodium hydrogen phosphate, sodium dihydrogen phosphate per injection.The routine of administration is Intramuscular injection into deltoid region.And the immunization schedule is two doses of quadrivalent influenza vaccine on day 0, 28.
  Arms: Control Group of trivalent influenza vaccine(BV)
Biological: Trivalent influenza vaccine(BY) — 7.5μg inactivated influenza antigen (H1N1, H3N2, and Yamagata) of each of the trivalent influenza vaccine in 0.25 mL of sodium chloride, disodium hydrogen phosphate, sodium dihydrogen phosphate per injection.The routine of administration is Intramuscular injection into deltoid region.And the immunization schedule is two doses of quadrivalent influenza vaccine on day 0, 28.
  Arms: Control Group of trivalent influenza vaccine(BY)

SUMMARY:
The study of quadrivalent influenza vaccine manufactured by Sinovac Biotech Co., Ltd will conduct in two phases,the phaseⅠclinical trial of the study will be open-label design,and the phase III clinical trial of the study will be randomized, double-blind, active controlled design.the purpose of this study is to evaluate the safety and immunogenicity of quadrivalent influenza vaccine in healthy subjects aged 6 to 35 months.

DETAILED DESCRIPTION:
This study of quadrivalent influenza vaccine will be open-label design in phase Ⅰ and randomized, double-blind, active controlled design in phase III.The quadrivalent influenza vaccine was manufactured by Sinovac Biotech Co., Ltd.

The purpose of this study is to evaluate the safety and immunogenicity of quadrivalent influenza vaccine(0.25ml and 0.5ml) manufactured by Sinovac Biotech Co., Ltd in healthy infants aged from 6 to 35 months. A total of 3330 subjects including 30 subjects in phase Ⅰ and 3300 subjects in phase III will be enrolled. The subjects in phase Ⅰ will receive 2 doses of quadrivalent influenza vaccine(0.5ml) on the immunization schedule of day 0,28.The subjects in phase III will be randomly assigned to 4 groups in a 2:2:1:1 ratio and subjects will receive two doses of quadrivalent influenza vaccine(0.25ml or 0.5ml) or trivalent influenza vaccine(BV or BY), respectively,on the immunization schedule of day 0,28 in each group.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants aged 6-35 months;
* Proven vaccination certificate and birth certificate;
* The subjects' guardians can understand and voluntarily sign the informed consent form.

Exclusion Criteria:

* Received any circulating seasonal influenza vaccine prior to enrollment or had an influenza vaccine schedule during the study;
* Suffering from seasonal influenza in the past 6 moths;
* Axillary temperature >37.0°C;
* History of asthma, history of allergy to the vaccine or vaccine components, or serious adverse reactions to the vaccine, such as urticaria, dyspnea, and angioedema;
* Congenital malformations or developmental disorders, genetic defects, severe malnutrition, etc.;
* Severe chronic diseases(Such as down syndrome, diabetes, sickle cell anaemia or neurological disorders);
* Severe neurological disease (epilepsy, convulsions or convulsions) or mental illness;
* Autoimmune disease or immunodeficiency / immunosuppression;
* Thyroid disease or history of thyroidectomy, asplenia,functional asplenia, asplenia or splenectomy resulting from any condition;
* Diagnosed abnormal blood coagulation function (eg, lack of blood coagulation factors, blood coagulopathy, abnormal platelets) or obvious bruising or blood coagulation;
* Immunosuppressive therapy, cytotoxic therapy, inhaled corticosteroids (excluding allergic rhinitis corticosteroid spray therapy, acute noncomplicated dermatitis superficial corticosteroid therapy) in the past 6 months;
* Acute diseases or acute exacerbation of chronic diseases in the past 3 days;
* Receipt of blood products within in the past 3 months;
* Receipt of other investigational drugs in the past 30 days;
* Receipt of attenuated live vaccines in the past 14 days;
* Receipt of inactivated or subunit vaccines in the past 7 days;
* Participated in other clinical trials before enrollment and in the follow-up period, or plans to participate in other clinical trials during the clinical trial;
* According to the investigator's judgment, the subject has any other factors that are not suitable for participating in the clinical trial

Ages: 6 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 217 (Actual)
Dates: Start 2022-08-08 (Actual); Primary Completion 2023-08-04 (Actual); Study Completion 2023-08-04 (Actual)

PRIMARY OUTCOMES:
Immunogenicity index of seroconversion rate | 28 days after full schedule immunization
  HI antibody seroconversion rate 28 days after full schedule immunization
Immunogenicity index of seroprotection rate | 28 days after full schedule immunization
  HI antibody seroprotection rate 28 days after full schedule immunization
Immunogenicity index of GMT | 28 days after full schedule immunization
  HI antibody GMT increase folds 28 days after full schedule immunization
Safety index of the incidence of adverse reaction | 0-28 days after each dose
  Incidence of adverse reaction 0-28 days after each dose
Safety index of the incidence of adverse reaction | 0-7 days after each dose
  Incidence of adverse reaction 0-7 days after each dose
Safety index of the incidence of abnormal blood biochemical indexes | 3 days after each dose
  The incidence of abnormal blood biochemical indexes 3 days after each dose
Safety index of the incidence of SAE | Since the beginning of vaccination until 6 months after full course vaccination
  Incidence of SAE since the beginning of vaccination until 6 months after full course vaccination

SECONDARY OUTCOMES:
Safety index of the incidence of AESI | Since the beginning of vaccination until 6 months after full course vaccination
  Incidence of AESI since the beginning of vaccination until 6 months after full course vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Hongxing Pan, Master, Principal Investigator — Jiangsu Provincial Center for Disease Prevention and Control
Locations (4):
- China (4):
  - Huaiyin Center for Diseases Control and Prevention, Huai'an, Jiangsu
  - Ganyu District Center for Disease Control and Prevention, Lianyungang, Jiangsu
  - Donghai District Center for Disease Prevention and Control, Lianyungang, Jiangsu
  - Binhai District Center for Disease Control and Prevention, Yancheng, Jiangsu